CLINICAL TRIAL: NCT05241223
Title: An Online Behavior Change Intervention to Promote Physical Activity in Adults With Asthma: a Randomized Controlled Trial
Brief Title: An Online Behavior Change Intervention to Promote Physical Activity in Adults With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Norte do Paraná (Other)
Responsible Party: Principal Investigator, Karina Furlanetto, Professor, Universidade Norte do Paraná
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OliveiraJM_PhD_FurlanettoKC
Record Dates: First submitted 2022-01-22; First posted 2022-02-15 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Asthma; Sedentary Behavior; Physical Inactivity
MeSH Terms: conditions — Asthma; Sedentary Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Sham Comparator): This group will receive an education program which will cover information regarding asthma, physical activity and sedentary behavior.
  Interventions: Other: Educational program
- Experimental group (Experimental): In addition to the educational program, this group will receive weekly individual and/or group online sessions for 12 weeks of motivation-based on behavior change intervention to promote physical activity and reduce sedentary behavior, based on both self-determination theory and transtheoretical model. They will also receive a pedometer with specific strategies related to it.
  Interventions: Other: Behavior change intervention

INTERVENTIONS:
Other: Behavior change intervention — This is an online intervention based on the transtheoretical model, along with self-determination theory strategies. This intervention will take place weekly summing up 12 online individual and/or group sessions of approximately 20 minutes. The sessions will be made through a platform and/or application that makes video calls privately. Each session will address a topic. In addition, in all sessions, the patients gain during the previous week will be recognized, as well as new goals will be set for the next week. The goals will always be individualized, realistic and achievable, based on the identification of each person's capacity and motivation. A Fitbit Zip will be used to propose objective goals aimed at increasing physical activity and reduce sedentary behavior. Additionally, a complex practice environment will be created around this device, such as the visualization of the number of steps evolution and competitions/games with other participants, among others.
  Arms: Experimental group
Other: Educational program — The educational program will be delivered similarly to both groups through videos and booklets, which will be sent in all weekdays during de first week after the initial assessment. Later, one educational material will be sent every two weeks until de 11th week. In the first day, patients will receive a quick welcome video call, in which information will be provided on how this program will work. In the subsequent days, the material will be sent daily and the participants will be able to ask questions, if they want to. The program will cover information regarding the respiratory system, pathophysiology of asthma, asthma treatment, prevention strategies and medication instructions. It will also be briefly addressed the subjects: understanding physical activity and sedentarism, as well as the importance and benefits of being physically active and less sedentary.
  Arms: Control group

SUMMARY:
The aims of this study are to investigate the effectiveness of an online behavior change (BC) intervention in increasing physical activity (PA) and reducing sedentary behavior in adults with asthma, as well as, in improving other clinical outcomes, in short and medium term. In this single-blind randomized clinical trial, patients with clinically stable moderate to severe asthma, who are physically inactive and do not have cardiovascular and/or osteoneuromuscular impairments will be randomized into control (CG) or intervention (IG) groups (23 in each group). Both groups will carry out a minimum educational program. Additionally, the IG will receive weekly individual and/or group online sessions for 12 weeks of motivation-based BC intervention to promote PA and reduce sedentary behavior, based on both self-determination theory (SDT) and transtheoretical model (TTM). The IG will also receive a pedometer with specific strategies related to it. Both groups will be reassessed immediately after the intervention as well as 6 months after the end of the intervention. The primary outcomes are PA and sedentary behavior, which will be objectively assessed by a triaxial accelerometer (Actigraph wGT3X-BT). Secondary outcomes are: asthma control, functional capacity, quality of life, sleep quality and symptoms of anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* people aged from 18 to 60 years
* diagnosis of moderate to severe asthma, who underwent drug treatment for at least 6 months
* clinical stability for at least 1 month (without hospitalizations, emergency care use or medication changes)
* absence of cardiovascular and/or osteoneuromuscular diseases that could interfere/hinder the performance of tests and physical activity
* absence of lung diseases other than asthma
* preserved cognitive function
* non-smokers or ex-smokers with <10 pack-years
* report being physically inactive in accordance with current physical activity guidelines
* able to make video calls through any platform and/or free app available

Exclusion Criteria:

* presence of any new orthopedic limitation that hinders the performance of physical activity during the study
* perform ≥150 minutes per week of moderate to vigorous physical activity during the initial assessment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Time spent in physical activity | 12 weeks from randomization
  Time spent (in minutes and percentage of the day) in light-intensity and moderate to vigorous physical activities, measured by a triaxial activity monitor.
Number of steps per day | 12 weeks from randomization
  Number of steps per day measured by a triaxial activity monitor
Time spent in sedentary behavior | 12 weeks from randomization
  Time spent (in minutes and percentage of the day) in sedentary activities, measured by a triaxial activity monitor.

SECONDARY OUTCOMES:
Time spent in physical activity | 36 weeks from randomization
  Time spent (in minutes and percentage of the day) in light-intensity and moderate to vigorous physical activities, measured by a triaxial activity monitor.
Number of steps per day | 36 weeks from randomization
  Number of steps per day measured by a triaxial activity monitor.
Time spent in sedentary behavior | 36 weeks from randomization
  Time spent (in minutes and percentage of the day) in sedentary activities, measured by a triaxial activity monitor.
Asthma control | 12 weeks from randomization
  Asthma Control Questionnaire score ranging from 0 to 6; the lower, the better.
Asthma control | 36 weeks from randomization
  Asthma Control Questionnaire score ranging from 0 to 6; the lower, the better.
Asthma symptoms and exacerbations | 12 weeks from randomization
  Frequency of asthma symptoms and exacerbations
Asthma symptoms and exacerbations | 36 weeks from randomization
  Frequency of asthma symptoms and exacerbations
Asthma medication use | 12 weeks from randomization
  Frequency of asthma rescue medication use
Asthma medication use | 36 weeks from randomization
  Frequency of asthma rescue medication use
Incremental Step Test | 12 weeks from randomization
  Number of steps climbed; the more the better
Incremental Step Test | 36 weeks from randomization
  Number of steps climbed; the more the better
Sit-To-Stand test | 12 weeks from randomization
  Number of repetitions in 1 minute; the more the better
Sit-To-Stand test | 36 weeks from randomization
  Number of repetitions in 1 minute; the more the better
Timed Up-and-Go test | 12 weeks from randomization
  Time to perform the test; the faster the better
Timed Up-and-Go test | 36 weeks from randomization
  Time to perform the test; the faster the better
4-Metre Gait Speed test | 12 weeks from randomization
  Time to perform the test; the faster the better
4-Metre Gait Speed test | 36 weeks from randomization
  Time to perform the test; the faster the better
Quality of life score | 12 weeks from randomization
  Asthma Quality of Life Questionnaire; ranges from 1 to 7 points; the higher the score, the better the quality of life
Quality of life score | 36 weeks from randomization
  Asthma Quality of Life Questionnaire; ranges from 1 to 7 points; the higher the score, the better the quality of life
Sleep quality | 12 weeks from randomization
  Subjectively measured by Pittsburgh Sleep Quality Index (score ranges from 0 to 21; the lower, the better) and objectively measured by Actiwatch 2 (Philips Respironics, Murrysville, Pennsylvania, USA).
Sleep quality | 36 weeks from randomization
  Subjectively measured by Pittsburgh Sleep Quality Index (score ranges from 0 to 21; the lower, the better) and objectively measured by Actiwatch 2 (Philips Respironics, Murrysville, Pennsylvania, USA).
Anxiety and depression symptoms | 12 weeks from randomization
  Hospital Anxiety and Depression Scale; ranges from 0 to 21 points; the higher the score, the worse the anxiety and depression symptoms
Anxiety and depression symptoms | 36 weeks from randomization
  Hospital Anxiety and Depression Scale; ranges from 0 to 21 points; the higher the score, the worse the anxiety and depression symptoms
Basic psychological needs | 12 weeks from randomization
  Basic Psychological Needs in Exercise Scale; ranges from 4 to 20; higher scores indicate greater levels of satisfaction of basic psychological needs
Basic psychological needs | 36 weeks from randomization
  Basic Psychological Needs in Exercise Scale; ranges from 4 to 20; higher scores indicate greater levels of satisfaction of basic psychological needs
Motivational regulations | 12 weeks from randomization
  Behavioral Regulation in Exercise Questionnaire; ranges from 0 to 4; the higher the score, the more regulated the individual is for a given level
Motivational regulations | 36 weeks from randomization
  Behavioral Regulation in Exercise Questionnaire; ranges from 0 to 4; the higher the score, the more regulated the individual is for a given level
Lung function | 12 weeks from randomization
  Spirometry determining the forced expiratory volume in the first second (FEV1), forced vital capacity (FVC) and FEV1/FVC index.
Lung function | 36 weeks from randomization
  Spirometry determining the forced expiratory volume in the first second (FEV1), forced vital capacity (FVC) and FEV1/FVC index.

CONTACTS AND LOCATIONS:
Overall Officials: Joice Oliveira, Msc, Principal Investigator — Universidade Norte do Paraná
Locations (1):
- Centro de Pesquisa e Pós Graduação na Unopar, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Oliveira JM, Pedroso A, de Melo DIF, Cunha MCA, de Lima FF, Carvalho CRF, Karloh M, Matias TS, Furlanetto KC. Short and medium term efficacy of an online behaviour change intervention on physical activity in adults with asthma. Sci Rep. 2026 Jan 8;16(1):4272. doi: 10.1038/s41598-025-34470-w. PMID 41501383
- [Derived] de Oliveira JM, Karloh M, Matias TS, Barbosa GB, Freitas PD, Carvalho CRF, Furlanetto KC. An online behavior change intervention to promote physical activity in adults with asthma: study protocol for a multicenter randomized controlled trial. Trials. 2022 Dec 7;23(1):983. doi: 10.1186/s13063-022-06881-x. PMID 36476386